CLINICAL TRIAL: NCT06899997
Title: Exploring the Effects of Time-restricted Feeding on the Immune Function of Obese Individuals: Multi-omic Approach
Brief Title: Study of the Effects of Time-Restricted Feeding on the Immune Function of Individuals With Obesity
Acronym: OBESIMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230714; 2023-A01185-40 (Other: Agence nationale de sécurité du médicament et des produits de santé); 24.04388.000237 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2025-03-13; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Obesity; Immune system
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Investigator aim to recruit a group of patients with obesity to test the effect of TRF on immune function and a group of patients with normal weight as a reference group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-restricted feeding (Experimental): Women with grade 3 obesity (BMI 40-50 kg/m²) who are scheduled for bariatric surgery and follow a time-restricted feeding (TRF) pattern consisting of an 8 h eating window (from 6-8 am to 14-16 pm) followed by a 16 h fasting period.
  Interventions: Other: Time-restrictred feeding
- Non-Time restricted feeding (Experimental): Women with grade 3 obesity (BMI 40-50 kg/m²) who are scheduled for bariatric surgery and follow a 14h eating window (from 6-8 am to 8-10 pm), followed by a 10 h fasting period.
  Interventions: Other: Non-time restricted feeding
- Control (No Intervention): Women with a healthy body weight without any dietary intervention

INTERVENTIONS:
Other: Time-restrictred feeding — Time-restricted feeding pattern consisting of an 8 h eating window (from 6-8 am to 14-16 pm) followed by a 16 h fasting period
  Arms: Time-restricted feeding
Other: Non-time restricted feeding — 14h eating window (from 6-8 am to 8-10 pm), followed by a 10 h fasting period
  Arms: Non-Time restricted feeding

SUMMARY:
The goal of this randomized trial is to: 1) investigate the immunological landscape of patients with obesity and conduct an in-depth functional characterization of their immune system; and 2) precisely define the effects of time-restricted feeding (TRF) on immune function in patients with obesity; 3) define the immunomodulatory properties of white adipocytes in response to TRF, and 4) uncover the underlying mechanisms by which TRF modulates the immune system patients with obesity through a multi-omics approach.

The main questions it aims to answer are: i) what is the underlying cause of impaired immunocompetence in patients with obesity? ii) how nutritional interventions improve the immune function of patients with obesity? Patients with obesity following TRF (8 h eating window ranging from 6-8 am to 14-16 pm) will be compared to patients with obesity without TRF control schedule (14h eating window ranging from 6-8 am to 8-10 pm). The dietary intervention will begin 10 weeks before the scheduled date for bariatric surgery in patients with obesity. In addition to patients with obesity, the present study aims to recruit a group of a reference healthy group (BMI between 18.5-24.9 kg/m²) that will not receive any nutritional intervention.

The following endpoints will be collected: Body weight and composition using Bioelectrical Impedance Analysis, resting energy expenditure (REE) using indirect calorimetry, blood glucose levels using a continuous glucose monitoring (CGM) device, metabolic parameters (fasting blood glucose levels, C-peptide, HbA1c, insulin, HOMA-IR, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, hepatic enzymes), and cytokine profile.

Blood, stool, and white adipose tissue (WAT) samples will be collected to establish metagenomic, transcriptomic, cytomic and metabolomic analyses.

ELIGIBILITY:
Inclusion Criteria:

Patients with obesity

* Women
* Age 18-64 years
* Body mass Index between 40-50 kg/m²
* Scheduled bariatric surgery 10-12 weeks after the nutritional intervention
* Self-reported eating pattern window of more than 14h
* Three meal eating pattern
* Stable body weight (less than 10% of current body weight during the last 3 months)
* Patients who have a favourable decision from the multidisciplinary team meetings after multidisciplinary nutritional follow-up of at least 6 months and history of failure with non-surgical weight loss methods
* Social security affiliation
* Written consent
* Good understanding of the French language

Lean patients

* Women
* Age 18-64 years
* Body mass Index between 18.5-24.9 kg/m²
* Scheduled banal surgery in the opinion of the investigator
* Self-reported eating pattern window of more than 14h
* Social security affiliation
* Written consent
* Good understanding of the French language

Exclusion Criteria:

* Diabetes type I or II
* Major cardiovascular disease
* Pregnancy
* Medication that could affect the study outcomes (i.e. anti-inflammatory drugs, antibiotics, immunosuppressors)
* Use products intended for weight loss
* Night work shift
* Past record of malignant tumors
* Serious liver dysfunction or chronic kidney disease
* Eating disorders
* Chronic viral disease (Hepatitis B or C, HIV) or inflammatory systemic diseases (i.e. Crohn's disease, rheumatoid arthritis)
* Serious cardiovascular or cerebrovascular disease within 6 months before randomization
* Severe gastrointestinal diseases or gastrointestinal surgery in the 12 months before randomization
* Under guardianship, curatorship, deprived of liberty
* Unable or unwilling to sign the informed consent form.
* Patient on AME (state medical aid)

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Level of inflammatory cytokine IL-1β | 10 weeks
  The mean difference in inflammatory cytokine IL-1β in patients with obesity after 10 weeks under TRF versus patients with obesity without TRF.

SECONDARY OUTCOMES:
Percent of weight change from baseline | Baseline, Week 10
Change in lean mass (expressed in kg), measured using Bioelectrical Impedance Analysis from baseline | Baseline, Week 10
Change in fat mass (expressed in kg), measured using Bioelectrical Impedance Analysis from baseline | Baseline, Week 10
Change in resting energy expenditure (kcal/day), measured using indirect calorimetry, from baseline | Baseline, 10 weeks
Change in fasting blood glucose levels from baseline | Baseline, 10 weeks
Change in fasting C-peptide levels from baseline | Baseline, 10 weeks
Change in HbA1c Levels from Baseline (Percentage Points) | Baseline, 10 weeks
Change in fasting insulin levels from baseline | Baseline, 10 weeks
Change in HOMA-IR from baseline | Baseline, 10 weeks
Change in lipid profile from baseline | Baseline, 10 weeks
Change in ALT and AST levels (U/L) from baseline | Baseline, 10 weeks
Change in Plasma Cytokine Levels from Baseline Using Luminex Assay | Baseline, 10 weeks
Changes in blood metabolome evaluated by gas chromatography and liquid chromatography coupled with high-resolution mass spectrometry | Baseline, 10 weeks
Changes in gut microbiome diversity using shotgun metagenomics | Baseline, 10 weeks
Changes in adipose tissue metabolome | Baseline, 10 weeks
Changes in gene expression profile assessed by RNA sequencing | Baseline, 10 weeks
Changes in blood immune cell populations measured using spectral flow cytometry | Baseline, 10 weeks
Changes in adipose tissue immune cell populations | Baseline, 10 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HEGP - digestive surgery, Paris
  - HEGP - nutrition department, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).